CLINICAL TRIAL: NCT03209401
Title: Niraparib Plus Carboplatin in Patients With Homologous Recombination Deficient Advanced Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Georgetown University (Other)
Collaborators: Tesaro, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0085
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor, Adult; Homologous Recombination Deficiency
Keywords: Niraparib; Carboplatin
MeSH Terms: interventions — niraparib; Carboplatin

STUDY DESIGN:
Intervention Model Description: The Phase Ia portion of the trial will be conducted in a 3+3 design, enrolling patients in cohorts of 3 patients each to insure safety and tolerability.
  There will be a Phase Ib expansion cohort including 20 patients to further assess the efficacy of niraparib plus carboplatin, using the RP2D and schedule from Phase Ia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib and Carboplatin (Experimental): Niraparib will be administered orally, once daily for 21 days of each 21-day cycle in escalating doses depending on cohort patient is assigned to.
  Carboplatin will be administered via an injection on Day 2 of a given 21-day cycle. The dose a patient receives will depend on which cohort the patient is assigned to.
  Interventions: Drug: Niraparib; Drug: Carboplatin

INTERVENTIONS:
Drug: Niraparib — an oral PARP inhibitor
  Other Names: MK-4827
Drug: Carboplatin — a platinum-based injection
  Other Names: Paraplatin

SUMMARY:
This is a multi-institutional Phase I dose-escalation and dose-expansion trial for patients with advanced, solid tumor malignancies who have pre-identified deleterious germline or somatic mutations in the homologous recombination deoxyribonucleic acid (DNA) repair pathway (HR deficient). The trial is designed to assess the efficacy and safety of niraparib plus carboplatin in patients with evidence of HRD. The primary endpoint will be identifying the recommended phase 2 dose (RP2D) and schedule of niraparib plus carboplatin, as well as establishing the anti-tumor efficacy of niraparib plus carboplatin as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

DETAILED DESCRIPTION:
This is a multi-institutional Phase I dose-escalation and dose-expansion trial for patients with advanced, solid tumor malignancies who have pre-identified deleterious germline or somatic mutations in the homologous recombination deoxyribonucleic acid (DNA) repair pathway (HR deficient). The trial is designed to assess the efficacy and safety of niraparib plus carboplatin in patients with evidence of HRD. The primary endpoint will be identifying the recommended phase 2 dose (RP2D) and schedule of niraparib plus carboplatin, as well as establishing the anti-tumor efficacy of niraparib plus carboplatin as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

Patients will be pre-identified from participating centers as having either a germline deleterious mutation or tumor expression of a deleterious mutation in one of the genes listed below, as determined by Next-generation DNA sequencing (NGS) only, completed prior to enrollment in this protocol. Patients with advanced solid tumor malignancies with the presence of somatic or germline deleterious mutation in a gene(s) critical to DNA repair through homologous recombination, including but not limited to: ARID1A, ATM, ATRX, MRE11A, NBN, PTEN, RAD50/51/51B, BARD1, BLM, BRCA1, BRCA2, BRIP1, FANCA/C/D2/E/F/G/L, PALB2, WRN, CHEK2, CHEK1, BAP1, FAM175A, SLX4, MLL2 or XRCC, and who have an adequate performance status (PS), bone marrow, hepatic, and renal function as well as biopsiable and measurable disease will be screened for enrollment.

Appropriate patients will be enrolled in a 3+3 alternating dose escalating fashion, to a maximum dose of niraparib of 300mg daily and a maximum dose of carboplatin area under the curve (AUC) of 4. The 3+3 schema will be employed to insure safety and tolerability. However, within any given cohort, a full contingent of 6 patients (assuming adequate tolerability) will be enrolled to capture a sufficient number of patients and samples for pharmacodynamic assessment of DNA damage.

Once the RP2D and schedule are identified, a Phase Ib expansion cohort of 20 additional patients will be enrolled as a pilot subgroup to determine efficacy. Of the 20 patients in this Phase Ib cohort, no more than 10 patients will have underlying breast cancer; and additionally no more than 10 patients may harbor BRCA1 or BRCA2 mutations.

To assess the efficacy of poly (ADP-ribose) polymerase (PARP) inhibition and the extent of DNA damage, patients will undergo serial tumor biopsies to measure DNA damage as quantified by levels of ᵞH2AX and RAD51 foci formation, as well as an assessment of PARP inhibitory activity. Tumor biopsies will also be used to assess the mechanisms of resistance to PARP inhibitor-based therapy.

Assessment of safety including blood tests, clinic visits and exams will occur weekly at the start of therapy, then will transition to every 3-week clinic visits and exams at the beginning of cycle 4. For the Phase Ib portion, patients will undergo weekly lab work and clinic visits for cycle 1 only. The researchers hypothesize that in this HR deficient patient population, the addition of niraparib to carboplatin will lead to significant anti-tumor responses with acceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients PRE-identified as having either a germline deleterious mutation or tumor expression of a deleterious mutation) as determined by Next-generation DNA sequencing only, in at least one gene involved in DNA damage repair through homologous recombination including but not limited to: ARID1A, ATM, ATRX, MRE11A, NBN, PTEN, RAD50/51/51B, BARD1, BLM, BRCA1, BRCA2, BRIP1, FANCA/C/D2/E/F/G/L, PALB2, WRN, CHEK2, CHEK1, BAP1, FAM175A, SLX4, MLL2 or XRCC.
* Patients with somatic mutations will be PRE-identified as having a homologous recombination mutation based on NGS done in a CLIA certified, CAP tested and bioinformatics-validated testing lab PRIOR to enrollment in this current protocol. The testing may have been done at any time prior to enrollment. HOWEVER, if any patient has had NGS testing more than 3 months prior to enrollment, or if there has been intervening therapy, then a repeat NGS test must be done and the deleterious somatic mutation must be re-identified for inclusion.
* The determination of a deleterious mutation must be supported in the documentation included in the testing, and should include clinical, or pre-clinical literature to support the finding that a specific mutation results in impaired function of the gene, and thus impaired DNA repair through homologous recombination. Variants of unknown significance will not be eligible.
* Patients with germline deleterious mutations may have been identified at any time point prior to inclusion in the protocol and do NOT need to have this genetic testing repeated regardless of time frame and intervening therapy.
* Advanced, solid tumor malignancy that is amenable to biopsy. Patient must consent to 4 mandatory biopsies during study
* Life expectancy of more than 3 months
* Age ≥ 18 years
* Measurable disease by RECIST v1.1 criteria (tumor ≥ 1 cm in longest diameter on axial image on computed tomography (CT) or magnetic resonance imaging (MRI) and/or lymph node(s) ≥ 1.5 cm in short axis on CT or MRI) on baseline imaging
* ECOG performance status (PS) of 0 to 1 (Table 10, Appendix A)
* Patients who have received and failed, or have been intolerant to, standard first line therapies known to confer clinical benefit. Patients who refuse standard therapy would also be eligible, as long as their refusal is documented.
* Patients with a standard 12-lead electrocardiogram (ECG) with the following parameters at screening (defined as the mean of the triplicate ECGs):

  1. QTc interval at screening < 481 msec
  2. Resting heart rate 50-90bpm
* Adequate hepatic, bone marrow, and renal function at the time of enrollment:
* Bone Marrow: Absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 9.0 g/dL. Patients must be able to meet the criteria without transfusion or receipt of colony stimulating factors within 2 weeks before obtaining sample
* Renal function: Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 50 mL/min/1.73 m2
* Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × the upper normal limit of institution's normal range. Total bilirubin ≤ 1.5 × the upper normal limit of institution's normal range. For subjects with liver metastases, AST and ALT < 5 × the upper normal limit of institution's normal range, and total bilirubin >1.5 - 3.0 x the upper normal limit of institution's normal range are acceptable as long as there is no persistent nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia
* Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) must be ≤ 2 X the upper limit of the institution's normal range and International Normalized Ratio (INR) < 2.

Subjects on anticoagulation (such as coumadin) will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator

* Patients may have received an unlimited number of prior therapies
* Patients must have fully recovered from all effects of surgery. Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring conscious sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patient is capable of swallowing pills whole
* Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the IRB, prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

* Prior disease progression while receiving platinum chemotherapy or platinum chemotherapy within the last 6 months
* For patients who received platinum-based adjuvant chemotherapy, at least 6 months must have passed between the last dose of platinum-based therapy and the development of metastatic disease. For breast cancer patients, at least 12 months must have passed between the last dose of platinum-based therapy and the development of metastatic disease
* Prior PARP inhibitor-based therapy
* Known or suspected CNS metastases, unless at least one month has passed since last local CNS therapy and there is no evidence for recurrent or progressive CNS disease on follow up imaging. Participants may remain on steroids for CNS disease if they are taking a stable dose
* Active severe infection, or known chronic infection with HIV or hepatitis B virus (testing not required prior to enrollment)
* Patients with chronic Hepatitis C virus may be enrolled if there is no clinical/laboratory evidence of cirrhosis AND the patient's liver function tests fall within the parameters set in Section 3.2.8.3, Inclusion Criteria, Hepatic function
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months. Additionally, patients must not have QT prolongation greater than or equal to 481 milliseconds
* Life-threatening visceral disease or other severe concurrent disease that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Presence of a psychiatric illness or social situation that would limit compliance with study requirements
* Women who are pregnant or breastfeeding
* The subject must not have had diagnosis, detection, or treatment of another type of cancer ≤2 years prior to randomization (except basal or squamous cell carcinoma of the skin that has been definitively treated). Questions regarding the inclusion of individual subjects should be directed to the Principal Investigators, Dr. Isaacs and Dr. Pishvaian.
* Clinically significant peripheral neuropathy at the time of enrollment (defined in the NCI CTCAE v4.0) as grade 2 or greater neurosensory or neuromotor toxicity)
* Patients must not have had investigational therapy administered ≤4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study
* Patients must not have had radiotherapy encompassing >20% of the bone marrow
* Patients must not have a known hypersensitivity to the components of niraparib or the excipients
* Patients must not have had any known, persistent > Grade 2 toxicity from prior cancer therapy
* Patient must not have had any known, persistent (>4 weeks), ≥Grade 3 hematological toxicity or fatigue from prior cancer therapy
* Patients must not have current evidence of any condition, therapy, or laboratory abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study or interfere with the patient's participation for the full duration of the study treatment or that makes it not in the best interest of the patient to participate
* Patients must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Patient must not have any known history of myelodysplastic syndrome (MDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Grade 3 and 4 toxicities | 36 months
  Phase Ia Primary Endpoint - The number of grade 3 and 4 toxicities according to NCI CTCAE; Version 4.0 that occur after Cycle 1, Day 1 will be recorded at each study visit.
Anti-tumor efficacy by overall response rate | 36 months
  Phase Ib Primary Endpoint - ORR is defined as the proportion of patients whose best overall response recorded during the treatment is either complete response or partial response according to the RECIST v1.1.

SECONDARY OUTCOMES:
Median survival | 36 months
  OS is defined by time from study enrollment till death from any cause
Median progression free survival | 36 months
  PFS is defined as the time from study enrollment to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first
Disease control rate | 36 months
  DCR is defined as the proportion of patients with a documented CR, PR, or SD at 4 months according to the RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT03209401/Prot_SAP_000.pdf